CLINICAL TRIAL: NCT00991952
Title: A Multicenter Random Assignment Phase II Study of Irinotecan and Alvocidib (Flavopiridol) Versus Irinotecan Alone for Patients With p53 Wild Type Gastric Adenocarcinoma
Brief Title: Irinotecan Hydrochloride With or Without Alvocidib in Treating Patients With Advanced Stomach or Gastroesophageal Junction Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-03825; NCI-2011-03825 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000655636; MSKCC-8060; 8060; 09-074 (Other: Memorial Sloan-Kettering Cancer Center); 8060 (Other: CTEP); N01CM00038 (NIH)
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2014-01-21 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2013-12

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gastric Cancer; Stage IIIC Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — alvocidib; Irinotecan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A (irinotecan hydrochloride, alvocidib) (Experimental): Patients receive irinotecan hydrochloride IV over 30 minutes and alvocidib IV over 1 hour on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Drug: irinotecan hydrochloride; Other: laboratory biomarker analysis
- Arm B (irinotecan hydrochloride) (Active Comparator): Patients receive irinotecan hydrochloride as in Arm A. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
  Arms: Arm A (irinotecan hydrochloride, alvocidib)
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well giving irinotecan hydrochloride with or without alvocidib works in treating patients with advanced stomach or gastroesophageal junction cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Alvocidib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether irinotecan hydrochloride is more effective with or without alvocidib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the antitumor efficacy of irinotecan (irinotecan hydrochloride) followed by flavopiridol (alvocidib) (Arm A) and of irinotecan alone (Arm B) in patients with advanced gastric/ gastroesophageal junction (GEJ) adenocarcinoma wild type for p53.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity of both study arms in patients with advanced gastric/GEJ adenocarcinoma.

II. To examine other measures of antitumor activity in both study arms, including response rate (in patients with measurable disease) and overall survival.

TERTIARY OBJECTIVES:

I. To evaluate pre- and post-treatment tumor biopsies for p21 and RAD51 homolog (S. cerevisiae) (Rad51) expression in patients who agree to tumor biopsies (Memorial Sloan-Kettering Cancer Center [MSKCC] and Weill-Cornell only).

II. To explore the response to irinotecan and flavopiridol and to irinotecan alone by deoxyribonucleic acid (DNA) microarray technology on pre- and post-treatment tumor biopsies (MSKCC and Weill-Cornell only).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive irinotecan hydrochloride intravenously (IV) over 30 minutes and alvocidib IV over 1 hour on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive irinotecan hydrochloride as in Arm A. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have pathologically confirmed carcinoma of the stomach or GEJ (Siewert's type I, II, or III); confirmation will be performed locally at each participating institution
* The patient must have advanced disease not amenable to surgical resection
* Patients must have disease that can be evaluated radiographically; this may be measurable disease or non-measurable disease; measurable disease is defined as that which can be measured in at least one dimension as > 20 mm with conventional techniques, or > 10 mm by high resolution imaging; disease that is identified on radiology studies, but does not meet the criteria for measurable disease, is considered non-measurable
* The patient must have received one prior chemotherapy regimen for his or her unresectable or metastatic disease; this does not include therapy administered in the adjuvant or neoadjuvant setting
* At least 2 weeks must have elapsed since the patient received prior chemotherapy, anti-angiogenic therapy, or other targeted therapy; 2 weeks since prior radiation therapy; or, 4 weeks if the last regimen included carmustine (BCNU) or mitomycin C
* The patient must have a Karnofsky performance status of >= 60
* Serum creatinine =< 2 mg/dl
* Total serum bilirubin =< 2 mg/dl

  * If the patient has Gilbert's disease and has a serum bilirubin greater than 2.0 mg/dl, the case must be discussed with the principal investigator; such a patient may be considered eligible on a case-by-case basis
* Serum aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 times the upper limit of normal, or
* Serum AST (SGOT)/ ALT (SGPT) =< 5 times the upper limit of normal in case of liver metastases
* White blood cell (WBC) >= 3000/mm^3
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelets >= 75,000/mm^3
* The patient must have available tumor tissue for assessment of p53 status by immunohistochemistry (IHC) (=< 20% cutoff for positivity)
* Tumor must be p53 wild type as defined as =< %20 nuclear staining on immunohistochemistry
* Women of child-bearing potential and sexually active males must be counseled to use an accepted and effective method of contraception (including intrauterine device [IUD], oral contraceptives, or barrier devices) while on treatment and for at least two months after their last treatment on this study; woman also must agree to refrain from nursing during the duration of this study and for at least two months after their last treatment on this study; women of child-bearing potential must have a negative serum pregnancy test to be eligible for this study
* The patient must have the mental capacity to understand the nature of this study and provide informed consent to participate

Exclusion Criteria:

* The patient may not have previously received irinotecan or flavopiridol
* The patient may not be receiving any other investigational agents
* The patient may not have any ongoing grade 2 or greater toxicity from a prior treatment
* The patient may not have an ongoing uncontrolled illness including, but not limited to active infection, symptomatic congestive heart failure, myocardial infarction in the past 6 months, or new cardiac arrhythmia in the past 6 months
* Patients with a diagnosis of active human immunodeficiency virus (HIV) infection, on anti-retroviral therapy, or with a cluster of differentiation 4 (CD4) count less than 200 are ineligible due to potential interactions between irinotecan, flavopiridol, and anti-retroviral medications as well as possible immunosuppressive activity of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 09/09/2009 Protocol Closed to Accrual 02/28/2012 Recruitment Location is the medical clinic
Groups:
- Irinotecan Hydrochloride and Alvocidib: Patients receive irinotecan hydrochloride IV over 30 minutes and alvocidib IV over 1 hour on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Irinotecan: 100 mg/m2 IV over 30 min on days 1 and 8 followed 7 hours later by Flavopiridol 60 mg/m2 IV over 1 hr on days 1 and 8
- Irinotecan Hydrochloride: Patients receive irinotecan hydrochloride as in Arm A. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Irinotecan: 100 mg/m2 IV over 30 min on days 1 and 8
Period: Overall Study
Arm/Group | Irinotecan Hydrochloride and Alvocidib | Irinotecan Hydrochloride
Started | 13 | 6
Completed | 13 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irinotecan Hydrochloride and Alvocidib | Irinotecan Hydrochloride | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (19.0918830) | 56 (16.97056275) | 60 (22.627417)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response was determined as indicated in the protocol.
Time Frame: From the start of treatment for up to 3 months
Measure: Number; unit: participants
Arm/Group | Irinotecan Hydrochloride and Alvocidib | Irinotecan Hydrochloride
Number analyzed (Participants) | 13 | 5
participants
  Partial Response | 1 | 0
  Stable Disease | 4 | 1
  Progression of Disease | 8 | 4

ADVERSE EVENTS:
Arm/Group | Irinotecan Hydrochloride and Alvocidib | Irinotecan Hydrochloride
Serious Adverse Events (participants affected / at risk) | 6/13 | 2/6
Other Adverse Events (participants affected / at risk) | 13/13 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan Hydrochloride and Alvocidib (N=13) | Irinotecan Hydrochloride (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Death-Disease Progression NOS (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decrease (Investigations) | 1 (1) | 0 (0)
Obstruction, gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan Hydrochloride and Alvocidib (N=13) | Irinotecan Hydrochloride (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (4) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Aspartate aminotransferase (Investigations) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (9) | 3 (3)
Fever (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (9) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
INR increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Neutrophil count decreased (Investigations) | 6 (6) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Weight loss (Investigations) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 10 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less